CLINICAL TRIAL: NCT06853210
Title: Treatment of Pressure Ulcers Using Biological Skin Substitutes: A Comparison of High Purity Type-I Collagen and Amnion/Chorion Membranes
Brief Title: Treatment of Pressure Ulcers Using Biological Skin Substitutes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adichunchanagiri Institute of Medical Sciences, B G Nagara (Other)
Responsible Party: Principal Investigator, Dr Naveen Narayan MS, MCh (Plastic Surgery), Professor and HOD, Adichunchanagiri Institute of Medical Sciences, B G Nagara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIMS/IEC/012/2025
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Pressure Sore
Keywords: Pressure Sore; High Purity Type I Collagen; Helicoll; Biological Skin Substitute; Dehydrated Human Amnion/Chorion Membrane
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High Purity Type-I Collagen-based Skin Substitute (Active Comparator): The SOC in this study is wound care covering with High Purity Type-I Collagen-based Skin Substitute applied weekly or as needed followed by a padded 3-layer dressing
  Interventions: Device: Type-I Collagen-based Skin Substitute and SOC
- Dehydrated Human Amnion/Chorion Membrane (Active Comparator): The SOC in this study is wound care covering with Dehydrated Human Amnion/Chorion Membrane followed by a padded 3-layer dressing
  Interventions: Device: Human Amnion/Chorion Membrane and SOC

INTERVENTIONS:
Device: Type-I Collagen-based Skin Substitute and SOC — The SOC in this study is wound care covering with High Purity Type-I Collagen-based Skin Substitute applied weekly or as needed followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous, second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap
  Arms: High Purity Type-I Collagen-based Skin Substitute
Device: Human Amnion/Chorion Membrane and SOC — The SOC in this study is wound care covering with Dehydrated Human Amnion/Chorion Membrane followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous, second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap
  Arms: Dehydrated Human Amnion/Chorion Membrane

SUMMARY:
Pressure ulcers, also known as decubitus ulcers or bedsores, are localized injuries to the skin and underlying tissue resulting from prolonged pressure. Management of pressure sores is crucial due to their association with increased morbidity, healthcare costs, and reduced quality of life. This study aims to evaluate the efficacy of two treatment modalities: Type-I Collagen-based Skin Substitute (HPTC) vs. Dehydrated Human Amnion/Chorion Membrane (dHCAM)

DETAILED DESCRIPTION:
Pressure ulcers, also known as decubitus ulcers or bedsores, are localized injuries to the skin and underlying tissue resulting from prolonged pressure. They are prevalent in individuals with limited mobility, such as the elderly and those with spinal cord injuries, particularly in long-term care settings. Effective management of pressure ulcers is crucial to prevent complications and improve patient outcomes, includes pressure relief, wound care, and advanced therapies such as bioengineered skin substitutes. Management of pressure sores is crucial due to their association with increased morbidity, healthcare costs, and reduced quality of life. This study aims to evaluate the efficacy of two treatment modalities: Type-I Collagen-based Skin Substitute (HPTC) vs. Dehydrated Human Amnion/Chorion Membrane (dHCAM) in promoting the healing of pressure ulcers. While both products are used in wound management, direct comparative studies evaluating their efficacy in treating pressure ulcers are limited.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age or older
2. Presence of a Stage II or Stage III pressure ulcer, as defined by the National Pressure Ulcer Advisory Panel
3. Ulcer size between 5 cm² and 25 cm²
4. Ulcer duration of at least 4 weeks prior to enrollment
5. The subject must agree to attend the twice-weekly/weekly study visits required by the protocol
6. The subject must be willing and able to participate in the informed consent process
7. Adequate blood supply to the affected area, confirmed by clinical assessment

Exclusion Criteria:

1. A subject known to have a life expectancy of <6 months
2. Presence of infection in the ulcer requiring systemic antibiotics.
3. Known allergy to components of HPTC or dHCAM.
4. Participation in another wound care study within the last 30 days.
5. A subject with autoimmune or connective tissue disorders.
6. Women who are pregnant or considering becoming pregnant within the next 6 months and those who are breast feeding.
7. History of autoimmune disease, immunosuppressive therapy, malignancy, or uncontrolled diabetes (HbA1c >10%)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prema Dhanraj, MS, MCh, Study Chair — Rajarajeshwari Medical College and Hospital
Locations (1):
- Adichunchanagiri Institute of Medical Sciences, Mandya, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergstrom N, Horn SD, Rapp MP, Stern A, Barrett R, Watkiss M. Turning for Ulcer ReductioN: a multisite randomized clinical trial in nursing homes. J Am Geriatr Soc. 2013 Oct;61(10):1705-13. doi: 10.1111/jgs.12440. Epub 2013 Sep 19. PMID 24050454
- [Background] Vecin NM, Kirsner RS. Skin substitutes as treatment for chronic wounds: current and future directions. Front Med (Lausanne). 2023 Aug 29;10:1154567. doi: 10.3389/fmed.2023.1154567. eCollection 2023. PMID 37711741
- [Background] Berhane CC, Brantley K, Williams S, Sutton E, Kappy C. An evaluation of dehydrated human amnion/chorion membrane allografts for pressure ulcer treatment: a case series. J Wound Care. 2019 May 1;28(Sup5):S4-S10. doi: 10.12968/jowc.2019.28.Sup5.S4. PMID 31067170
- [Background] Narayan N, Gowda S, Shivannaiah C. A Randomized Controlled Clinical Trial Comparing the Use of High Purity Type-I Collagen-Based Skin Substitute vs. Dehydrated Human Amnion/Chorion Membrane in the Treatment of Diabetic Foot Ulcers. Cureus. 2024 Dec 5;16(12):e75182. doi: 10.7759/cureus.75182. eCollection 2024 Dec. PMID 39649230

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 19 | 41
  >=65 years | 18 | 21 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 30
  Male | 28 | 22 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  India | 40 | 40 | 80
Ulcer duration [Mean (Standard Deviation); unit: Months] | 2.1 (1.1) | 2.3 (1.2) | 2.2 (1.15)
Ulcer size [Mean (Standard Deviation); unit: square centimeters] | 14.9 (2.1) | 15.0 (1.8) | 14.95 (1.94)
Ulcer Location Distribution [Count of Participants; unit: Participants]
  Gluteal region | 16 | 16 | 32
  Sacral region | 11 | 12 | 23
  Lateral malleolus | 5 | 6 | 11
  Heel | 6 | 4 | 10
  Elbow | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Wound Area
Description: Percent Change in Wound Area from week 1 through week 7 measured manually with digital photography
Time Frame: 7 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
percentage change | -78.5 (18.2) | -65.1 (9.8)

2. Primary Outcome: Histopathological Parameters - Vascular Infiltration
Description: A 2mm punch biopsy was obtained from the wound edge extending into the wound bed under local anaesthesia. Serial sections of 4μm thickness were prepared and stained with Hematoxylin and Eosin (H&E) for general morphology.
  Vascular Infiltration: Assessed by counting new blood vessels per High Power Field (hpf) (0-3 scale) 0: Minimal vascular ingrowth (<5 vessels/hpf)
  1. Mild infiltration (5-10 vessels/hpf)
  2. Moderate infiltration (11-20 vessels/hpf)
  3. Abundant infiltration (>20 vessels/hpf) (0-worse; 3-better)
Time Frame: Baseline (Day 0), Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
Participants
  Day 0 / Baseline: Grade 0 | 11 | 17
  Day 0 / Baseline: Grade 1 | 15 | 14
  Day 0 / Baseline: Grade 2 | 8 | 6
  Day 0 / Baseline: Grade 3 | 6 | 3
  Day 5 Post Application: Grade 0 | 0 | 4
  Day 5 Post Application: Grade 1 | 2 | 13
  Day 5 Post Application: Grade 2 | 7 | 15
  Day 5 Post Application: Grade 3 | 31 | 8

3. Primary Outcome: Histopathological Parameters - Neo-epithelialization
Description: A 2mm punch biopsy was obtained from the wound edge extending into the wound bed under local anaesthesia. Serial sections of 4μm thickness were prepared and stained with: Hematoxylin and Eosin (H&E) for general morphology. Neo-epithelialization: Measured as epithelial migration distance from wound edge (0-3 scale) 0: No epithelial migration
  1. Minimal migration (<25% wound coverage)
  2. Moderate migration (25-75% coverage)
  3. Extensive migration (>75% coverage) (0-worse; 3-better)
Time Frame: Baseline (Day 0), Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
Participants
  Day 0 / Baseline: Grade 0 | 18 | 24
  Day 0 / Baseline: Grade 1 | 12 | 10
  Day 0 / Baseline: Grade 2 | 7 | 4
  Day 0 / Baseline: Grade 3 | 3 | 2
  Day 5 of Post Application: Grade 0 | 0 | 6
  Day 5 of Post Application: Grade 1 | 4 | 15
  Day 5 of Post Application: Grade 2 | 8 | 10
  Day 5 of Post Application: Grade 3 | 28 | 9

4. Primary Outcome: Histopathological Parameters - Fibroblast Activity
Description: A 2mm punch biopsy was obtained from the wound edge extending into the wound bed under local anaesthesia. Serial sections of 4μm thickness were prepared and stained with: α-SMA immunohistochemistry for fibroblast activity. Fibroblast Activity: Quantified by counting α-SMA positive fibroblasts per HPF and assessment of fibroblast morphology (0-3 scale) 0: Sparse, inactive fibroblasts
  1. Moderate cellularity, minimal matrix production
  2. High cellularity, active-matrix synthesis
  3. Very high activity with extensive matrix deposition (0-worse; 3-better)
Time Frame: Baseline (Day 0), Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
Participants
  Day 0 / Baseline: Grade 0 | 7 | 12
  Day 0 / Baseline: Grade 1 | 17 | 16
  Day 0 / Baseline: Grade 2 | 13 | 10
  Day 0 / Baseline: Grade 3 | 3 | 2
  Day 5 Post Application: Grade 0 | 0 | 3
  Day 5 Post Application: Grade 1 | 2 | 15
  Day 5 Post Application: Grade 2 | 5 | 15
  Day 5 Post Application: Grade 3 | 33 | 7

5. Primary Outcome: Histopathological Parameters - Inflammatory Response
Description: 2mm punch biopsy was obtained from the wound edge extending into the wound bed under local anaesthesia.
  Serial sections of 4μm thickness were prepared and stained with: Hematoxylin and Eosin (H&E) for general morphology Inflammatory Response: Graded semi-quantitatively (0-3 scale) 0: Minimal inflammatory infiltrate
  1. Mild chronic inflammation
  2. Moderate mixed inflammation
  3. Severe acute inflammation
  (0-better; 3-worse)
Time Frame: Baseline (Day 0), Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
Participants
  Day 0 / Baseline: Grade 0 | 21 | 12
  Day 0 / Baseline: Grade 1 | 14 | 16
  Day 0 / Baseline: Grade 2 | 5 | 11
  Day 0 / Baseline: Grade 3 | 0 | 1
  Day 5 Post Application: Grade 0 | 20 | 9
  Day 5 Post Application: Grade 1 | 17 | 12
  Day 5 Post Application: Grade 2 | 3 | 15
  Day 5 Post Application: Grade 3 | 0 | 4

6. Primary Outcome: Histopathological Parameters - Capillary Density
Description: A 2mm punch biopsy was obtained from the wound edge extending into the wound bed under local anaesthesia.
  Serial sections of 4μm thickness were prepared and stained with: CD31 immunohistochemistry for capillary density evaluation Capillary Density: Evaluated using CD31 staining, counted as vessels per mm² of tissue
  More the vessels per square centimeters better
Time Frame: Baseline (Day 0), Day 5
Measure: Mean (Standard Deviation); unit: vessels per square centimeters
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
vessels per square centimeters | 47.3 (8.2) | 28.7 (9.6)

7. Primary Outcome: Histopathological Parameters - Collagen Deposition
Description: A 2mm punch biopsy was obtained from the wound edge extending into the wound bed under local anaesthesia. Serial sections of 4μm thickness were prepared and stained with: Masson's Trichrome for collagen assessment Collagen Deposition: Assessed using Masson's Trichrome staining (0-3 scale) 0: Minimal collagen matrix
  1. Loose, immature collagen
  2. Moderate organized collagen
  3. Dense, mature collagen architecture
  (0-worse; 3-better)
Time Frame: Baseline (Day 0), Day 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
score on a scale | 2.63 (0.49) | 1.77 (0.63)

8. Secondary Outcome: Complete Wound Closure Rates
Description: Percentage of subjects to obtain complete closure, defined as 100% epithelialization with no drainage, of the target ulcer was determined by the proportion of subjects that obtain complete closure over the 6-week treatment period and additional 1 week follow up
Time Frame: 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
Participants | 30 | 25

9. Secondary Outcome: Wound Size Progression Over Time
Description: Mean wound sizes at each time point for both treatment groups assessing change in wound size throughout the study period. Assessed from baseline, through day 5, 14th day, 21 st day, 28th, 35th and 42nd days of HPTC or dHACM application
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: sqauare centimeters
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
sqauare centimeters
  Baseline | 14.9 (2.1) | 15.0 (1.8)
  Day 5 | 13.1 (2.3) | 13.4 (2.1)
  Day 14 | 11.1 (2.4) | 11.5 (2.2)
  Day 21 | 9.1 (2.8) | 9.8 (2.1)
  Day 28 | 7.0 (3.1) | 8.2 (2.4)
  Day 35 | 5.2 (3.2) | 6.8 (2.6)
  Day 42 | 3.2 (3.1) | 5.2 (2.4)

10. Secondary Outcome: Mean Number of Repeated Application
Description: Mean number of reapplications of the HPTC & dHACM used to obtain wound closure over 6 Weeks
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mean number of reapplications
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
mean number of reapplications | 0.85 (0.92) | 1.15 (0.87)

11. Secondary Outcome: Adverse Events
Description: Adverse events (e.g., infection, allergic reactions)
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
Participants
  No adverse event | 38 | 34
  Mild Erythema | 2 | 4
  Mild Allergic Reaction | 0 | 2
  Severe adverse events | 0 | 0

12. Secondary Outcome: Patient Treatment Satisfaction
Description: Patient treatment satisfaction will be assessed by using a validated 5-point Likert scale questionnaire administered at 7 weeks post-treatment initiation. The questionnaire evaluated overall treatment satisfaction, comfort during application, perceived effectiveness, and willingness to recommend the treatment to others, measured with score range from 1 to 5, wherein 1="Extremally Unsatisfied" to 5="Extremally Satisfied"
Time Frame: 7 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
score on a scale | 4.33 (0.62) | 3.41 (0.78)

13. Other Pre Specified Outcome: Change in Quality of Life
Description: Change in quality of life assessed using the Wound-QoL questionnaire measured as 'not at all', 'a little', 'moderately', 'quite a lot' and 'very much' for 17 questions and total number of patients who reported improvement in Quality of Life was measured
Time Frame: 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
Number analyzed (Participants) | 40 | 40
Participants
  Improvement | 29 | 17
  No Change | 11 | 19
  Worsening | 0 | 4

ADVERSE EVENTS:
Time Frame: 7 weeks
Description: All the study participants were considered at risk for adverse events.
Arm/Group | High Purity Type-I Collagen-based Skin Substitute | Dehydrated Human Amnion/Chorion Membrane
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 2/40 | 6/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Purity Type-I Collagen-based Skin Substitute (N=40) | Dehydrated Human Amnion/Chorion Membrane (N=40)
Mild Erythema (Immune system disorders) | 2 (2) | 4 (4)
Mild Allergic Reaction (Immune system disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Single-centre design may limit generalizability to other healthcare settings and populations.

Relatively short follow-up period (7 weeks), while sufficient for assessing acute healing outcomes, may not capture long-term outcomes, recurrence rates or durability of treatment effects.

The Study was not completely blinded due to the nature of the interventions Study included a specific range of wound sizes and may not be generalizable to very large wounds.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT06853210/Prot_SAP_001.pdf